CLINICAL TRIAL: NCT05731934
Title: A Phase I Clinical Trial of the Tolerability and Pharmacokinetics of HX301 Monolactate Capsules in Patients With Advanced Solid Tumors
Brief Title: The Tolerability and Pharmacokinetics of HX301 Monolactate Capsules in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Hanx Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX301-I-01
Record Dates: First submitted 2023-01-29; First posted 2023-02-16 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HX301 (Experimental): Study treatment: during each cycle (28 days), HX301 is dosed QD for 3 weeks (21 days) followed by 1 week (7 days) off therapy.
  Interventions: Drug: HX301

INTERVENTIONS:
Drug: HX301 — At starting dose of 40 mg, followed by 4 dose levels of 80 mg, 120 mg, 160 mg, and 200 mg
  Other Names: HX301 Monolactate Capsules

SUMMARY:
Open label, single- and multiple-dose administration, dose-exploratory clinical phase I study to evaluate the safety, tolerability and PK profile of HX301 monolactate capsules in patients with advanced malignant solid tumors and to preliminarily evaluate its antitumor efficacy.

DETAILED DESCRIPTION:
The study is divided into a screening period (28 days before first dose), treatment period, and follow-up period.

In the dose escalation stage, the study will follow a 3+3 dose-escalation scheme enrolling cohorts of at least 3 subjects sequentially at escalating doses. The dose escalation phase includes a single-dose phase and a multiple-dose phase. Subjects in the single-dose phase were treated with HX301monolactate, taken orally before breakfast, and in the multiple-dose phase, the frequency of administration was once daily (QD), 3 weeks continuously, suspended for 1 week, and every 4 weeks (28 days) was a dosing cycle. Dose escalation will continue until identification of an MTD or the maximum dose is reached. Dose-limiting toxicities (DLTs) will be assessed from the first dose of study treatment until 28 days. Blood samples will be collected at regular intervals for pharmacokinetics (PK).

The Tumor evaluation (assessed by the Investigator in accordance with Response Evaluation Criteria in Solid Tumors Version 1.1 [RECIST 1.1] to assess efficacy will start from the first dose and occur every 8 weeks in the first 24 weeks and every 12 weeks thereafter.

After 1 year of treatment, if the sponsor and investigator determine that the subject can still benefit from treatment with HX301, the treatment may continue until the disease progresses, the investigator determines that the subject is no longer suitable for further treatment, the subject voluntarily withdraws from the treatment, or the sponsor withdraws the trial.

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntarily agree to sign informed consent, understand the study and is willing and able to comply with all the trial procedures.

  2) Male or female subject aged 18-75 years (including the boundary value). 3) Patients with cytologically or histopathological confirmed advanced malignant solid tumors that is refractory/relapsed to standard therapy (with disease progression or intolerance) or lack of effective treatment, or the subject refuses standard therapy.

  4) Eastern Cooperative Oncology Group performance status of 0 to 1. 5) Life expectancy at least 3 months. 6) Subjects with measurable lesions (at least 1 extracranial lesion) according to the solid tumor evaluation criteria (RECIST v1.1).

  7) For subjects who have received prior anti-tumor therapy, as follows:
  * Systemic radiotherapy ≥ 3 weeks before the first dose, local radiotherapy to bone metastasis ≥ 2 weeks prior to the first administration of study treatment.
  * Previous chemotherapy, immunotherapy (PD-1 antibody, PD-L1 antibody or CTLA-4 antibody, etc.), biological anti-tumor therapy (tumor vaccine, cytokines or growth factors), and targeted therapy ≥ 4 weeks before the first dose (small molecule targeted therapy ≥ 2 weeks prior to the first dose).
  * Previously received anti-tumor herbal medicine or medications which content herbal ingredient approved for anticancer, with an interval of ≥ 2 weeks prior to the first dose.

    8) Subjects may have a history of brain/meningeal metastases, provided they have received local treatment (including surgery and radiotherapy, etc.) and have been stable for at least 3 months prior to the first dose.

    9) Adequate organ and bone marrow hematopoietic function, as evidenced by:
* Absolute neutrophil count (ANC) ≥ 1.5×109/L.
* absolute white blood cell count (WBC) ≥ 3.0×109/L.
* Platelet count ≥ 100×109/L.
* Hemoglobin ≥ 90 g/L (not treated with blood transfusion within 2 weeks before the first dose)
* Serum creatinine ≤ 1.5 1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min (calculated according to the Cockcroft-Gault formula, see Annex 6)
* Serum total bilirubin (TBIL) ≤1.5 x upper limit of normal (ULN).
* AST and ALT ≤ 2.5 x ULN, and ≤ 5 x ULN in subject with liver cancer or liver metastases.
* International normalized ratio (INR) ≤ 2 x ULN or activated partial thromboplastin time (APTT) ≤ 1.5 x ULN (unless the subject is on anticoagulation therapy, then as long as the PT or APTT is within the expected therapeutic range for anticoagulant use).

  10) Male subjects and female subjects of childbearing potential should agree to use effective contraception from the time they sign the informed consent until 3 months after the last dose.

Exclusion Criteria:

* Subjects are excluded from the study if any of the following criteria apply:

  1. Patients with other malignant tumors within 5 years before enrollment, except cured cervical carcinoma in situ and cured cutaneous basal cell carcinoma.
  2. Failure to recover from previously treated adverse reactions to CTCAE 5.0 grade ≤ 1, except for residual alopecia effects.
  3. previous use or ongoing use of antitumor agents targeting CDK4/6
  4. inability to swallow, chronic diarrhea and intestinal obstruction with multiple factors affecting drug uptake and absorption
  5. Planning major surgery (excluding diagnostic surgical procedures) during this study including the 28-day screening period
  6. The presence of uncorrectable hypokalemia and hypomagnesemia found to remain during the screening period.
  7. Presence of third interstitial fluid that cannot be controlled by drainage or other means (e.g., massive pleural fluid, ascites, pelvic effusion).
  8. uncontrolled and stable systemic diseases, such as severe hypertension, diabetes mellitus, thyroid disease, etc.
  9. unstable angina pectoris, myocardial infarction, or heart failure within 3 months prior to the first dose of the drug; a history of a heart rate disorder requiring drug treatment or considered clinically significant by the investigator; any other cardiac disease considered by the investigator to be inappropriate for participation in this trial, etc.; and cardiac function abnormalities of ≥ grade II severity (according to NYHA classification, see Annex 7) found during the screening period examination.
  10. History of infection with human immunodeficiency virus, or other acquired, congenital immunodeficiency diseases, or history of organ transplantation, or history of stem cell transplantation.
  11. Patients with active chronic hepatitis B or active hepatitis C or active syphilis, hepatitis B virus carriers, patients with stable hepatitis B after drug treatment (DNA titer < 500 IU/mL or DNA copy number <103 copies/mL), cured hepatitis C patients (HCV RNA test negative) and cured syphilis patients (syphilis antigen negative ) can be enrolled.
  12. Those with severe infections within 4 weeks before the first dose.
  13. Participation in other drug clinical trials within 4 weeks prior to the first dose.
  14. Patients with a clear history of neurological or psychiatric disorders, such as epilepsy, dementia, and poor compliance.
  15. Female subject who is pregnant or lactating.
  16. Subjects who, per the opinion of the investigator, are not suitable for participation in this trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) in HX301 Monolactate Capsules in patients with advanced solid tumors | Collected adverse events from first dosing through at least 30 days after the end of treatment, or until other cancer treatment regimens have been started (whichever occurs earlier)
  Adverse events (AEs) determined by the investigator are recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0).
Incidence of Dose Limiting Toxicities (DLT) in HX301 Monolactate Capsules in patients with advanced solid tumors | 7 days after single dose (C0D1-C0D7) and 4 weeks after first dose of multiple dose (C1D1-C1D28).
  Incidence of Dose Limiting Toxicities (DLT) that would result in stopping dosing

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum plasma concentration of drug (Cmax) | Single dose : Cycle 0 Day 1 and multiple dose : Cycle 1 Day 1,Cycle 1 Day 8,Cycle 1 Day 9,Cycle 1 Day 15 (each cycle is 28 days)
  Highest concentration of drug measured in the PK samples
Pharmacokinetics(PK): Time to reach Cmax (Tmax) | Single dose : Cycle 0 Day 1 and multiple dose : Cycle 1 Day 1,Cycle 1 Day 8,Cycle 1 Day 9,Cycle 1 Day 15 (each cycle is 28 days)
  Time from dosing until collection of the PK samples with the highest drug concentration.
Terminal Half-life （t½）of HX301 | Single dose : Cycle 0 Day 1 and multiple dose : Cycle 1 Day 1,Cycle 1 Day 8,Cycle 1 Day 9,Cycle 1 Day 15 (each cycle is 28 days)
  Terminal phase elimination half-life
Area Under the Serum Concentration-time Curve (AUC) | Single dose : Cycle 0 Day 1 and multiple dose : Cycle 1 Day 1,Cycle 1 Day 8,Cycle 1 Day 9,Cycle 1 Day 15 (each cycle is 28 days)
  The area under the serum concentration-time curve .
Objective response rate (ORR) of HX301 Monolactate Capsules in patients with solid tumors | Approximately 1 years
  The ORR is defined as the percentage of participants in the analysis population who had a confirmed Complete Response or Partial Response.
Duration of response (DoR) of HX301 Monolactate Capsules in patients with solid tumors | Approximately 1 years
  The DoR is defined as the time from the first recorded response (CR or PR) to the first recorded tumor progression or death due to any cause.
Progression-free survival (PFS) of patients with solid tumors treated with HX301 | Approximately 1 years
  The PFS is defined as the time from the start of the first dose to the first documented disease progression or death of any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- National center/cancer hospital,chinese Academy of Medical Sciences and Peking Union Medicial College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No